CLINICAL TRIAL: NCT03469882
Title: High Protein Intake and Early Exercise in Adult Intensive Care Patients: Impact on Functional Outcomes. A Randomized Controlled Phase II Trial.
Brief Title: High Protein Intake and Early Exercise in Adult Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, MD; PhD, Hospital Sao Domingos
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ICUHSD 03/18
Record Dates: First submitted 2018-03-11; First posted 2018-03-19 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Critically Ill Patients
Keywords: Protein, exercise, critical illness, outcome,
MeSH Terms: conditions — Motor Activity; Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinded outcomes assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein and exercise (HPE) group (Experimental): Begining within 48 hours of ICU admission participants will receive nutrition support with energy expenditure measured by indirect calorimetry, 2.0 to 2.2 g/kg/day of protein and in-bed cycle ergometry exercise.
  Interventions: Dietary Supplement: High protein nutrition; Device: Cycle ergometry exercise
- Usual care group (Other): Participants randomized to the usual care group will receive usual care protein and exercise
  Interventions: Other: Usual care group

INTERVENTIONS:
Dietary Supplement: High protein nutrition — Patients in the HPE group will be submitted to nutritional support preferably through the enteral route. Energy expenditure will be determined by indirect calorimetry. They will receive 2.0 to 2.2 grams/kg/day of protein.
  Arms: High protein and exercise (HPE) group
Device: Cycle ergometry exercise — Patients will be submitted to two daily sessions of exercise (cycle ergometry) 15 minutes duration each, during the 7 days of the week. The intervention will be maintained exclusively duting the patient's stay in the ICU. The cycle ergometer will be the MotoMed Letto II (Reck Technik, Germany).
  Arms: High protein and exercise (HPE) group
Other: Usual care group — Participants randomized to the usual care group will receive usual care protein and exercise.
  Other Names: No intervention
  Arms: Usual care group

SUMMARY:
This study analyse the impact of high protein intake associated to early programed exercise on functional outcomes of adult intensive care patients.

DETAILED DESCRIPTION:
The muscle weakness associated to intensive care, one of the components of Post Intensive Care Syndrome (PICS) has a significant impact on the short-term and long-term outcomes in the critically ill patient (1, 2). Puthucheary et al. (3) analyzed 63 septic patients with imaging examination and established a clear relationship between the number of organ failures and muscle loss in the first 10 days of ICU. Although a study involving 244 critically ill patients has shown an alarming relationship between reduced muscle mass at admission and mortality (4), evidences that nutritional interventions can attenuate muscle loss and result in improvement in outcome are unclear. Recent studies evaluating the impact of nutritional therapy on clinical outcomes have surprisingly demonstrated that patients who received full nutritional intake did not differ in outcomes when compared to those receiving reduced nutritional intake, the so-called permissive underfeeding (5, 6, 7). Careful analysis of these studies, however, reveals that the authors define hyponutrition as synonymous with reduced calorie intake, without mentioning the protein intake offered to the patients. The study with the greatest scientific repercussion (8) used reduced caloric intake in the study group, but the protein intake did not differ between groups. Observational studies comparing high protein intake with conventional intake have shown improvement in outcome indicators in patients receiving more than 1.6 and even more than 2.0 g / kg / day of protein (9, 10). Recently the intensive care medicine research agenda published in the journal of the European Society of Intensive Care Medicine, the top priority of the nutrition research in the critically ill patients was to compare normal and hyperproteic nutrition ideally associated with physical activity (11). Several recent studies have shown benefits of early physical rehabilitation in the critically ill patient (12, 13).

The optimal integration between adequate protein intake and exercise in the critically ill patient may have an impact on short- and long-term outcomes, but this hypothesis has not yet been tested by studies with a good methodology. The hypothesis of this prospective randomized phase II study is that the association of high protein intake with early physical rehabilitation improves physical function after hospital discharge with a significant impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

We will include 180 consecutive patients admitted to one of the study ICUs

* Aged 18 years or above.
* Non-pregnant.
* Requiring mechanical ventilation for at least 48 hours.
* Expected ICU stay higher than 3 days.

Exclusion Criteria:

* Inability to walk without assistance before the acute illness that led to ICU admission (use of gait aid is not an exclusion criterion).
* Cognitive impairment prior to hospitalization described by relatives and evaluated by the ICU psychology team.
* Neuromuscular diseases that compromise weaning from mechanical ventilation.
* Acute pelvic fracture.
* Unstable spinal cord trauma.
* Patients considered moribund.
* In some situations patients will not be included in the resistive exercise program for as long as a temporary limiting factor remains:
* Patients undergoing neuromuscular blocking drugs.
* Patients under high-dose vasoactive drug use.
* Mechanical ventilation with FIO2 (fraction of inspired oxygen) ≥ 60% and / or PEEP (positive end-expiratory pressure)> 12 cm H2O.
* Intracranial hypertension.
* . Open abdomen.
* Status epilepticus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Physical component summary (PCS) 3 months after randomization | 3 months after randomization
  Blind assessment of PCS after 3 months after randomization
Physical component summary (PCS) 6 months after randomization | 6 months after randomization
  Blind assessment of PCS after 6 months after randomization

SECONDARY OUTCOMES:
handgrip strength | 20 days
  handgrip strength measured at ICU discharge,
Duration of mechanical ventilation | 20 days
  Length of time under mechanical ventilation
Length of ICU stay | 20 days
  Length of ICU stay
Hospital mortality | 6 months
  Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: WIDLANI s MONTENEGRO, RN, Ms, Study Director — Hospital Sao Domingos
Locations (1):
- Icu Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Background] Doig GS, Simpson F, Sweetman EA, Finfer SR, Cooper DJ, Heighes PT, Davies AR, O'Leary M, Solano T, Peake S; Early PN Investigators of the ANZICS Clinical Trials Group. Early parenteral nutrition in critically ill patients with short-term relative contraindications to early enteral nutrition: a randomized controlled trial. JAMA. 2013 May 22;309(20):2130-8. doi: 10.1001/jama.2013.5124. PMID 23689848
- [Background] Harvey SE, Parrott F, Harrison DA, Bear DE, Segaran E, Beale R, Bellingan G, Leonard R, Mythen MG, Rowan KM; CALORIES Trial Investigators. Trial of the route of early nutritional support in critically ill adults. N Engl J Med. 2014 Oct 30;371(18):1673-84. doi: 10.1056/NEJMoa1409860. Epub 2014 Oct 1. PMID 25271389
- [Background] Arabi YM, Aldawood AS, Haddad SH, Al-Dorzi HM, Tamim HM, Jones G, Mehta S, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Afesh L; PermiT Trial Group. Permissive Underfeeding or Standard Enteral Feeding in Critically Ill Adults. N Engl J Med. 2015 Jun 18;372(25):2398-408. doi: 10.1056/NEJMoa1502826. Epub 2015 May 20. Erratum In: N Engl J Med. 2015 Sep 24;373(13):1281. doi: 10.1056/NEJMx150028. PMID 25992505
- [Background] Allingstrup MJ, Esmailzadeh N, Wilkens Knudsen A, Espersen K, Hartvig Jensen T, Wiis J, Perner A, Kondrup J. Provision of protein and energy in relation to measured requirements in intensive care patients. Clin Nutr. 2012 Aug;31(4):462-8. doi: 10.1016/j.clnu.2011.12.006. Epub 2011 Dec 29. PMID 22209678
- [Background] Nicolo M, Heyland DK, Chittams J, Sammarco T, Compher C. Clinical Outcomes Related to Protein Delivery in a Critically Ill Population: A Multicenter, Multinational Observation Study. JPEN J Parenter Enteral Nutr. 2016 Jan;40(1):45-51. doi: 10.1177/0148607115583675. Epub 2015 Apr 21. PMID 25900319
- [Background] Arabi YM, Casaer MP, Chapman M, Heyland DK, Ichai C, Marik PE, Martindale RG, McClave SA, Preiser JC, Reignier J, Rice TW, Van den Berghe G, van Zanten ARH, Weijs PJM. The intensive care medicine research agenda in nutrition and metabolism. Intensive Care Med. 2017 Sep;43(9):1239-1256. doi: 10.1007/s00134-017-4711-6. Epub 2017 Apr 3. PMID 28374096
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Background] Gruther W, Pieber K, Steiner I, Hein C, Hiesmayr JM, Paternostro-Sluga T. Can Early Rehabilitation on the General Ward After an Intensive Care Unit Stay Reduce Hospital Length of Stay in Survivors of Critical Illness?: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2017 Sep;96(9):607-615. doi: 10.1097/PHM.0000000000000718. PMID 28181920
- [Background] Chrispin PS, Scotton H, Rogers J, Lloyd D, Ridley SA. Short Form 36 in the intensive care unit: assessment of acceptability, reliability and validity of the questionnaire. Anaesthesia. 1997 Jan;52(1):15-23. doi: 10.1111/j.1365-2044.1997.015-az014.x. PMID 9014540
- [Background] Ciconelli RM, Ferraz MB, Santos W, Meirão 1, Quaresma MR. Brazilian-portuguese version of the SF-36. A reliable and valid quality of life outcome measure. Rev Bras Reumatologia. 1999; 39 (3): 143-50.
- [Derived] de Azevedo JRA, Lima HCM, Frota PHDB, Nogueira IROM, de Souza SC, Fernandes EAA, Cruz AM. High-protein intake and early exercise in adult intensive care patients: a prospective, randomized controlled trial to evaluate the impact on functional outcomes. BMC Anesthesiol. 2021 Nov 13;21(1):283. doi: 10.1186/s12871-021-01492-6. PMID 34773985